CLINICAL TRIAL: NCT04842786
Title: Topical Coconut Oil Application and Incidence of Sepsis in Neonates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Cloudnine Hospital, Bangalore, India (Unknown); University of Cincinnati (Other)
Responsible Party: Principal Investigator, Vivek Narendran, MD, Professor of Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-0487
Record Dates: First submitted 2021-04-02; First posted 2021-04-13 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Late-Onset Neonatal Sepsis
Keywords: late-onset neonatal sepsis; premature infant; full-term infant; skin; skin barrier; biomarker; stratum corneum; skin surface acidity (pH); transepidermal water loss; imaging; d'squame tape; microbiome; coconut oil
MeSH Terms: conditions — Neonatal Sepsis; Premature Birth | interventions — Coconut Oil

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, parallel group, controlled trial
Who Masked: Outcomes Assessor
Masking Description: Subjects will be randomly assigned to receive coconut oil or no treatment using a random number scheme after stratification for gestational age group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coconut oil at 5 mg/Kg body weight twice daily (Experimental): Coconut oil (Parachute Brand) is a marketed product that is routinely used for daily massage after birth for infants in India. An amount of 5 mg/Kg body weight will be applied twice daily by the health care provider from enrollment until discharge, or until day of life 28, whichever occurs first.
  Interventions: Other: Coconut oil
- No intervention (No Intervention): Subjects assigned to this arm will have their skin gently stroked twice daily for the time that would be required to apply an oil. This will simulate the stroking received by the intervention arm subjects. This will occur from enrollment until discharge, or until day of life 28, whichever occurs first.

INTERVENTIONS:
Other: Coconut oil — Coconut oil, Parachute oil composition: 92% lauric (C12) fatty acid, 6% oleic fatty acid, 2% linoleic fatty acid
  Arms: Coconut oil at 5 mg/Kg body weight twice daily

SUMMARY:
The randomized control trial aims to determine the effect of twice daily application of a commonly used coconut oil to the skin of neonates in the neonatal intensive care setting on the rate of late onset sepsis versus a no treatment control.

DETAILED DESCRIPTION:
Purpose and Specific Aims

The purpose is to determine the effect of twice daily topical coconut oil application on late onset sepsis in neonates admitted to the Neonatal Intensive Care Units of Indira Gandhi Institute of Child Health, Cloudnine Hospital at Old Airport Road, and Cloudnine Hospital at Jayanagar in Bangalore, India. The aim is to determine the effect of topical coconut oil application on:

* The incidence of neonatal late onset culture positive sepsis
* Neonatal skin integrity versus a no treatment control using standard skin evaluation methods
* Biomarkers of neonatal innate immune function
* Temperature instability, weight gain, intraventricular hemorrhage, necrotizing enterocolitis, retinopathy of prematurity, chronic lung disease, and mortality.

The investigators hypothesize that twice daily topical coconut oil application will reduce the incidence of late onset sepsis (LOS) in premature and full-term infants versus the current standard of care, i.e., no treatment. The oil treatment will increase the neonatal skin barrier integrity measured by validated clinical and instrumental methods. Skin surface biomarkers of innate immune function collected from coconut oil treated skin will indicate less inflammation (lower proinflammatory cytokine levels) than in untreated control skin.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants 24-36 weeks gestational age
* Full-term infants 37-42 weeks gestational age
* Less than 48 hours of age at enrollment
* Admitted to the neonatal intensive care unit of Indira Gandhi Institute for Child Health, Cloudnine Hospital at Old Airport Road and Cloudnine Hospital at Jayangar, Bangalore
* Expected to be in the neonatal intensive care unit for at least 4 days after enrollment
* Able to tolerate study procedures as described
* Parent/guardian willing to provide written informed consent

Exclusion Criteria:

* Medically unstable
* Parent/guardian unable to provide written informed consent
* Presence of inherited cutaneous condition e.g., scalded skin syndrome, epidermolysis bullosa
* Presence of major congenital anomalies
* Infants undergoing surgery

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Late-onset sepsis rate for intervention versus control | Day 3 of life until discharge or day of life 28, whichever occurs first
  Incidence of late-onset sepsis is defined as an infection that occurs on or after day 3 of life

SECONDARY OUTCOMES:
Skin erythema | Day 3 of life until discharge or day of life 28, whichever comes first
  The skin erythema (redness) of the outer thigh and perianal region will be quantified from visual inspection of high resolution digital photographs that will be collected with standard positioning and lighting and color corrected. The area of coverage and severity of erythema will be judged using published, validated grading scales.
Skin rash | Day 3 of life until discharge or day of life 28, whichever comes first
  The skin rash of the outer thigh and perianal region will be quantified from visual inspection of high resolution digital photographs that will be collected with standard positioning and lighting and color corrected. The area of coverage and severity of rash will be judged using published, validated grading scales.
Skin dryness | Day 3 of life until discharge or day of life 28, whichever comes first
  The skin dryness of the outer thigh and perianal region will be quantified from visual inspection of high resolution digital photographs that will be collected with standard positioning and lighting and color corrected. The area of coverage and severity of dryness/scaling will be judged using published, validated grading scales.
Skin transepidermal water loss | Day 3 of life until discharge or day of life 28, whichever comes first
  The rate of transepidermal water loss of a site on the outer thigh will be measured as grams/meter2/hour using a standard, closed-chamber instrument known as the Vapometer. This instrument will provide the transepidermal water loss value once the system reaches equilibrium. This method has previously been validated and is used routinely for skin measurements.
Skin surface acidity (pH) | Day 3 of life until discharge or day of life 28, whichever comes first
  The skin surface acidity of a site on the outer thigh and a site on the buttocks covered by the diaper will be measured using a flat surface electrode device that is calibrated daily to buffers of pH 4 and pH 7. The surface acidity is given in pH units which are the negative log to the base 10 of the hydrogen ion concentration of water placed on the skin by the instrument probe. The instrument is designed for use on the skin and has been validated.
Set of skin surface proteins of known innate immune function | Day 3 of life until discharge or day of life 28, whichever comes first
  There are proteins in the skin surface layers known to be biomarkers of innate immune function. Each protein will be quantified and reported as picograms of protein per microgram of total protein. The specific proteins are: filaggrin, filaggrin 2, transglutaminase 3, S100A8 (antimicrobial, calcium binding protein), S100A7 (antimicrobial, calcium binding protein), SERPINB3 (cysteine protease inhibitor), SERPINB4 (protease inhibitor), elafin (protease inhibitor) keratins 1, 6A and 6B (structural proteins) and fatty acid elongase 1 (lipid). Levels of each protein will be evaluated together to compare effect of the intervention versus control.
  Samples from skin surface will be collected using two sequential adhesive tapes (gentle adhesive) placed on the skin sites (thigh, buttocks covered by diaper) for one minute each, removed and stored at -80 deg C until analysis. The proteins will be extracted and analyzed for using standard techniques of tandem mass spectrometry.
Skin Microbiome | Day 3 of life until discharge or day of life 28, whichever comes first
  Microbiome analyses of neonatal skin and stool to determine the effect of coconut oil versus no treatment on microflora
Chronic lung disease | Day 3 of life until discharge or day of life 28, whichever comes first
  The incidence of chronic lung disease among the subjects in the intervention (coconut oil) will be compared to the incidence in the no treatment control during the study period. Chronic lung disease will be diagnosed based on the subject's oxygen requirement at 36 weeks corrected age.
Causative Organisms of Sepsis | Day 3 of life until discharge or day of life 28, whichever comes first
  Sepsis diagnosis includes determination of the organisms to which sepsis was attributed
Necrotizing enterocolitis | Day 3 of life until discharge or day of life 28, whichever comes first.
  The impact of coconut oil versus no treatment on the incidence of necrotizing enterocolitis during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Kumar, MBBS, MD, Principal Investigator — Cloudnine Hospital; Naveen Benakappa, MBBS, MD, Principal Investigator — Indira Gandhi Institute of Child Health; Prathik B H, MBBS, MD, Principal Investigator — Indira Gandhi Institute of Child Health
Locations (2):
- India (2):
  - Cloudnine Hospital, Bangalore
  - Indira Gandhi Institute of Child Health, Bangalore

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.